CLINICAL TRIAL: NCT05292443
Title: Therapeutic ResistAnce and Clonal Evolution Assessed With Liquid Biopsy in ICIs Treated Primary Liver Cancer
Status: Withdrawn | Type: Observational
Why Stopped: No participants were enrolled
Sponsor: Geneplus-Beijing Co. Ltd. (Industry)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HisPower-Lib 002
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Primary Liver Cancer; Hepatocellular Carcinoma; Intrahepatic Cholangiocarcinoma; Combined Hepatocellular-cholangiocarcinoma
Keywords: Next Generation Sequencing (NGS); Liquid biopsy; Immune Checkpoint Inhibitor; Whole Transcriptome Sequencing
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — whole blood (including plasma, white cells), tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — observe the association of ctDNA with efficacy of treatment

SUMMARY:
To evaluate the predictive value of ctDNA in response, relapse for liver cancer patients treated with immune checkpoint inhibitors

DETAILED DESCRIPTION:
In the study, 300 advanced primery liver cancer patients who received immune checkpoint inhibitors at first-line setting (N=200) or second-line setting (N=100) will be recruited. By analyzing the ctDNA and peripheral blood mononuclear cell (PBMC) collected before and after the first cycle of ICI treatment, the dynamic changes of bTMB, ctDNA and the composition of immune cells will be detected. Combined with the tumor markers AFP, DCP and CA19-9, a noninvasive multiparameter model will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Primary liver cancer diagnosed according to the clinical diagnostic criteria, or histopathological or cytological examination;
* 18-80 years old, no limit on gender;
* ECOG performance status of 0-2, with expected survival time of more than 12 weeks;
* According to RECIST V1.1, there must be at least one measurable lesion;
* Patients who are suitable for ICIs treatment and willing to comply with required protocols and give permission to use the data for clinical research and products development;
* Patients who join the study voluntarily, sign a consent form, have good compliance, and comply with follow-up.

Exclusion Criteria:

* Patients with other primary cancers;
* Patients with a severe parenchymal disease and unable to accept ICIs treatment;
* Patients with a psychiatric disorder and unable to comply with this study;
* Patients with symptomatic brain metastasis, anticipated complications or cognitive disorders that are associated with brain metastasis;
* Adverse events related to prior anti-tumor treatment (except for hair loss of any grade) did not return to grade 1 or better;
* History of cells or organ transplantation;
* History of hypersensitivity to the drug administered in this study or contrast media for CT and MRI;
* Patients who accepted hepatic local therapy (including ablation therapy, percutaneous injection of ethanol or acetic acid (PEI/PAI), high-intensity focused ultrasound (HIFU), transarterial chemoembolization (TACE)) within 14 days prior to initiation of the study;
* Other reasons that the researchers think not suitable for ICIs treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary liver cancer including hepatocellular carcinoma, intrahepatic cholangiocarcinoma and combined hepatocellular-cholangiocarcinoma
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
PFS: Progression-free survival | 24 months
  The time length from the date of randomization to any of the following events: disease progression or death from any cause.

SECONDARY OUTCOMES:
ORR: Objective Response Rate | 24 months
  The proportion of patients with complete response or partial response.
OS: Overall Survival | 24 months
  The time length from the date of randomization to the date of death.
TTD: Time to Treatment Discontinuation | 24 months
  The time length from the date of randomization to the date of treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, MD PhD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (5):
- China (5):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing hospital, Beijing, Beijing Municipality
  - Institute of Hepatopancreatobiliary Surgery, Chongqing General Hospital, University of Chinese Academy of Sciences (UCAS), Chongqing, Chongqing Municipality
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University, Wuhan, Hubei
  - Eastern Hepatobiliary Surgery Hospital, Second Military Medical University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided